CLINICAL TRIAL: NCT04562363
Title: Prevention of Postoperative Ventral Hernias After Median Laparotomy in Urgent Surgery
Brief Title: Prevention of Postoperative Ventral Hernias
Status: Completed | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: POVG12122021
Record Dates: First submitted 2020-08-28; First posted 2020-09-24 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2021-10

CONDITIONS: Gangrenous Postoperative Ventral Hernia (Diagnosis); Dehiscence of Laparotomy Wound
Keywords: Postoperative ventral hernia; eventrat; defects of the fascia; laparotomic wound suture; preventive prosthetics of a laparotomic wound
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low risk of herniation.: Use of any method of suturing, including modified.
  Interventions: Procedure: Suturing of a laparotomic wound with modified methods
- The average risk of hernia formation: The application of modified methods of closure of laparotomy wound.
  Interventions: Procedure: Suturing of a laparotomic wound with modified methods
- high risk of herniation: The use of alloplastic methods of closure of laparotomy wound.
  Interventions: Procedure: Suturing of a laparotomic wound with modified methods
- The presence of eventrations: The use of alloplastic methods of suturing a laparotomic wound in the absence of suppuration.
  Interventions: Procedure: Suturing of a laparotomic wound with modified methods

INTERVENTIONS:
Procedure: Suturing of a laparotomic wound with modified methods — Suturing the white line of the abdomen with the help of developed techniques aimed at preventing hernias and eventrations

SUMMARY:
The research is aimed at identifying factors of herniation after median laparotomy and developing surgical methods for preventing postoperative ventral hernias and eventrations.

DETAILED DESCRIPTION:
At the first stage, an analysis of the prevalence of postoperative ventral hernias in patients after median laparotomies in urgent surgery will be performed, with the identification of factors contributing to the development of postoperative ventral hernias. At the next stage, the investigators will search for the most reliable methods of suturing the white line of the abdomen, taking into account the risk of hernia formation, with their implementation in patients operated in an emergency through median laparotomic access in comparison with traditionally used methods. In conclusion, an algorithm will be developed for selecting the method of surgical prevention of postoperative ventral hernias, taking into account the risk of their development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes aged 18 years and older who are expected to perform median laparotomy on a planned or emergency basis.
2. Patients who have signed an informed consent to participate in the study, after the purpose and meaning of the study have been explained to them.
3. Patients who follow the doctor's instructions.

Exclusion Criteria:

1. The death of the patient.
2. Stage IV cancer
3. Hernia repair with hernioplasty, including simultaneous surgery
4. Refusal of the patient to cooperate with the researcher.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective study included 700 patients, including those operated through a midline laparotomic approach to identify factors of herniation, and those who are planned to have a midline laparotomy in order to choose a rational method of suturing a laparotomic wound, taking into account the risk of incisional hernia formation. Taking into account the degree of risk of postoperative ventral hernia development and the choice of the method of its prevention, the patients were divided into 4 groups.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Wound complications | 2 weeks
  Frequency of wound complications in the early postoperative period.
Eventration | 2 weeks
  Frequency of events in the early postoperative period
Pain syndrome | 2 year
  The severity of pain syndrome in the postoperative scar after midline laparotomy using a verbal scale of pain syndrome
Postoperative ventral hernia | 2 year
  Frequency of postoperative ventral hernia in the late postoperative period
Defects in the aponeurosis | 2 year
  Frequency of aponeurosis defects in the late postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Inyutin, PhD MD, Principal Investigator — RyazSMU
Locations (2):
- Russia (2):
  - RyazSMU, Ryazan, Ryazan Oblast
  - RyazSMU, Ryazan

IPD SHARING:
Plan to Share IPD: No
Undecided Basic demographic data, including sex, age, and ethnicity are to be shared if allowed by the privacy policy.